CLINICAL TRIAL: NCT02951455
Title: Community Wise: An Innovative Multi-level Intervention to Reduce Alcohol and Illegal Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Development and Research Institutes, Inc. (Other); University of Michigan (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); North Jersey Community Research Initiative (Other)
Responsible Party: Principal Investigator, Liliane Cambraia Windsor, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1U01MD010629-01 (NIH); 1U01MD010629-01 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- CD-LC (Experimental): Group behavioral intervention with 9 weekly sessions lasting 2 hours. Critical Dialogue (CD), Licensed Clinician (LC).
  Interventions: Behavioral: Critical Dialogue; Behavioral: LC
- CBP- LC (Experimental): Group community mobilizing intervention with 9 weekly sessions spread in 15 weeks. Capacity Building Project (CBP), Licensed Clinician (LC)
  Interventions: Behavioral: Capacity Building Project; Behavioral: LC
- QLW- LC (Experimental): Group intervention where participants learn to develop and implement personal goals that are measurable, attainable, realistic, and time bound. Intervention includes 9 sessions. Quality of Life Wheel, Licensed Clinician (LC)
  Interventions: Behavioral: Quality of Life Wheel; Behavioral: LC
- CD & CBP- LC (Experimental): Combination of group behavioral intervention and community mobilization intervention including 15 weekly sessions.Licensed Clinician (LC)
  Interventions: Behavioral: Critical Dialogue; Behavioral: Capacity Building Project; Behavioral: LC
- CD & QLW- LC (Experimental): Combination of group behavioral intervention and community mobilization intervention including 15 weekly sessions.Licensed Clinician (LC)
  Interventions: Behavioral: Critical Dialogue; Behavioral: Quality of Life Wheel; Behavioral: LC
- QLW & Capacity Building ProjectCBP- LC (Experimental): Combination of goal development and implementation with community mobilization intervention including 9 weekly sessions spread across 15 weeks. Licensed Clinician (LC)
  Interventions: Behavioral: Capacity Building Project; Behavioral: Quality of Life Wheel; Behavioral: LC
- QLW & CD & CBP-LC (Experimental): Combination of group behavioral intervention, goal development and implementation, and community mobilization intervention including 15 weekly sessions.Licensed Clinician (LC)
  Interventions: Behavioral: Critical Dialogue; Behavioral: Capacity Building Project; Behavioral: Quality of Life Wheel; Behavioral: LC
- LC (Experimental): This condition will include 3 core sessions that are not a part of the components being tested. These are support sessions to the components being tested and is hypothesized to have the smallest impact on substance use outcomes.Licensed Clinician (LC)
  Interventions: Behavioral: LC
- CD- PF (Experimental): Group behavioral intervention with 9 weekly sessions lasting 2 hours. Critical Dialogue (CD), Peer Facilitator (PF)
  Interventions: Behavioral: Critical Dialogue; Behavioral: PF
- CBP- PF (Experimental): Group community mobilizing intervention with 9 weekly sessions spread in 15 weeks. Capacity Building Project (CBP), Peer Facilitator (PF)
  Interventions: Behavioral: Capacity Building Project; Behavioral: PF
- QLW-PF (Experimental): Group intervention where participants learn to develop and implement personal goals that are measurable, attainable, realistic, and time bound. Intervention includes 9 sessions. Quality of Life wheel, Peer Facilitator (PF)
  Interventions: Behavioral: Quality of Life Wheel; Behavioral: PF
- CD & CBP- PF (Experimental): Combination of group behavioral intervention and community mobilization intervention including 15 weekly sessions. Peer Facilitator (PF)
  Interventions: Behavioral: Critical Dialogue; Behavioral: Capacity Building Project; Behavioral: PF
- CD & QLW- PF (Experimental): Combination of group behavioral intervention and community mobilization intervention including 15 weekly sessions.Peer Facilitator (PF)
  Interventions: Behavioral: Critical Dialogue; Behavioral: Quality of Life Wheel; Behavioral: PF
- QLW & CBP- PF (Experimental): Combination of goal development and implementation with community mobilization intervention including 9 weekly sessions spread across 15 weeks.Peer Facilitator (PF)
  Interventions: Behavioral: Capacity Building Project; Behavioral: Quality of Life Wheel; Behavioral: PF
- CD & QLW & CBP- PF (Experimental): Combination of group behavioral intervention, goal development and implementation, and community mobilization intervention including 15 weekly sessions.Peer Facilitator (PF)
  Interventions: Behavioral: Critical Dialogue; Behavioral: Capacity Building Project; Behavioral: Quality of Life Wheel; Behavioral: PF
- PF (Experimental): This condition will include 3 core sessions that are not a part of the components being tested. These are support sessions to the components being tested and is hypothesized to have the smallest impact on substance use outcomes. Peer Facilitator (PF)
  Interventions: Behavioral: PF

INTERVENTIONS:
Behavioral: Critical Dialogue — Prompted by thematic images, aims to help participants develop a deeper understanding of how marginalizing processes (e.g., systematic stigma; feelings of rage as victims of discrimination) impact participants' lives and behavior.
  Other Names: CD
  Arms: CD & CBP- LC; CD & CBP- PF; CD & QLW & CBP- PF; CD & QLW- LC; CD & QLW- PF; CD- PF; CD-LC; QLW & CD & CBP-LC
Behavioral: Capacity Building Project — Designed to create collaborative efforts to overcome and dismantle marginalizing processes by building positive social and organizational relationships and community capacity through the development and implementation of community projects aiming to address social determinants of health.
  Other Names: CBP
  Arms: CBP- LC; CBP- PF; CD & CBP- LC; CD & CBP- PF; CD & QLW & CBP- PF; QLW & CBP- PF; QLW & CD & CBP-LC; QLW & Capacity Building ProjectCBP- LC
Behavioral: Quality of Life Wheel — Aims to increase self-efficacy and help participants develop a vision for their future, breaking this vision down into small, feasible, measureable goals they can implement on a weekly basis (e.g. quitting smoking, improving relationships with family members, paying down debt).
  Other Names: QLW
  Arms: CD & QLW & CBP- PF; CD & QLW- LC; CD & QLW- PF; QLW & CBP- PF; QLW & CD & CBP-LC; QLW & Capacity Building ProjectCBP- LC; QLW- LC; QLW-PF
Behavioral: PF — Whether the intervention is delivered by a peer facilitator.
  Arms: CBP- PF; CD & CBP- PF; CD & QLW & CBP- PF; CD & QLW- PF; CD- PF; PF; QLW & CBP- PF; QLW-PF
Behavioral: LC — Whether the intervention is delivered by a licensed clinician.
  Arms: CBP- LC; CD & CBP- LC; CD & QLW- LC; CD-LC; LC; QLW & CD & CBP-LC; QLW & Capacity Building ProjectCBP- LC; QLW- LC

SUMMARY:
The current project seeks to implement the Multiphase Optimization Strategy (MOST) and Community Based Participatory Research (CBPR) principles to identify the most efficient, scalable, and sustainable combination of Community Wise components. Community Wise is a manualized multi-level intervention aimed at reducing health inequalities related to alcohol and illicit drug use (AIDU).This 2x2x2x2 factorial design will be fully powered to detect change in AIDU in a sample of 528 men with substance use disorders and a history of incarceration residing in distressed communities with predominantly Black populations. Participants will be randomly assigned to one of sixteen experimental conditions.

DETAILED DESCRIPTION:
The current project seeks to implement the Multiphase Optimization Strategy (MOST) and Community Based Participatory Research (CBPR) principles to identify the most efficient, scalable, and sustainable combination of Community Wise components. Community Wise is a manualized multi-level intervention aimed at reducing health inequalities related to alcohol and illicit drug use (AIDU). The research will be conducted by the Newark Community Collaborative Board (NCCB), a network that developed and pilot-tested the original Community Wise. NCCB members include the principal investigators (PIs), co-investigators (Co-Is), service providers, consumers of AIDU, and community members.

Specific aims include:

Aim 1: Use a highly efficient experimental design to estimate the unique contribution of key components of Community Wise in: a) reducing AIDU frequency and b) increasing the percentage of participants abstinent over five months. Components tested are the presence or absence of: (a) Critical Dialogue; (b) Quality-of-Life-Wheel; (c) Capacity Building Project; and (d) group facilitation by a peer versus a licensed clinician. A factorial experiment will be used to detect effects of individual components and three-way interactions.

Aim 2: Informed by MOST, Community Wise will be optimized for scalability and sustainability-- the most efficacious combination of components that can be delivered for less than $2000 per intervention cycle serving up to eleven individuals simultaneously (as per recommendations by the Substance Abuse and Mental Health Services Administration (SAMHSA).

This 2x2x2x2 factorial design will be fully powered to detect change in AIDU in a sample of 528 men with substance use disorders and a history of incarceration residing in distressed communities with predominantly Black populations. Participants will be randomly assigned to one of sixteen experimental conditions. The first eight conditions will be facilitated by a licensed facilitator. The remaining conditions will be facilitated by a peer facilitator. Each set of eight conditions will include the following components: (1) Critical Dialogue (CD) only; (2) Quality-of-Life-Wheel (QLW) only; (3) Capacity Building Project (CBP) only; (4) CD+QLW; (5) CD+CBP; (6) QLW+CBP; (7) CD+QLW+CBP; and (8) no components. Data will be collected at baseline plus five post-baseline monthly follow-ups. This study has potential to impact public health; the use of CBPR and MOST will generate action-oriented implications and an optimized multi-level intervention adaptable to address different health inequalities.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the factorial experiment participants in the study will include:

* Men age 18 or older
* Residence in Essex County, NJ
* Willingness to be voice recorded during group sessions
* Ability to speak English
* Having a substance use disorder measured by the Global Appraisal of Individual Needs-Substance Problem Scale (GAIN-SPS).
* Having been released from incarceration in the past 4 years. This is due to research that shows that people are more likely to be re-incarcerated within the first 4 years of release from incarceration.

Exclusion Criteria:

* Severe psychiatric disorders in the prior 6 months not stabilized (schizophrenia, depression with psychotic features, bipolar disorder, any psychosis), as measured by the MINI International Neuropsychiatric Interview 6 psychoticism and suicidality modules
* Gross cognitive impairment as measured by the Mini Mental State Exam.
* Sexual identification as female

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliane Windsor, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- Integrity House, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will require a data- sharing agreement that provides for the following conditions at minimum: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate tools and computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
  All data will be stripped of personal identifiers so as to be suitable for use by other investigators. Even though the database will be stripped of identifiers prior to any sharing, however, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for the above-stated commitments.

REFERENCES:
- [Derived] Windsor LC, Benoit E, Pinto RM, Gwadz M, Thompson W. Enhancing behavioral intervention science: using community-based participatory research principles with the multiphase optimization strategy. Transl Behav Med. 2021 Aug 13;11(8):1596-1605. doi: 10.1093/tbm/ibab032. PMID 33837786
- [Derived] Windsor LC, Benoit E, Smith D, Pinto RM, Kugler KC; Newark Community Collaborative Board (NCCB). Optimizing a community-engaged multi-level group intervention to reduce substance use: an application of the multiphase optimization strategy. Trials. 2018 Apr 27;19(1):255. doi: 10.1186/s13063-018-2624-5. PMID 29703237

RESULTS

PARTICIPANT FLOW:
Groups:
- Core LC: This condition will include 3 core sessions that are not a part of the components being tested. These are support sessions to the components being tested and is hypothesized to have the smallest impact on substance use outcomes.Licensed Clinician (LC)
  LC: Whether the intervention is delivered by a licensed clinician.
- Core PF: This condition will include 3 core sessions that are not a part of the components being tested. These are support sessions to the components being tested and is hypothesized to have the smallest impact on substance use outcomes. Peer Facilitator (PF)
  PF: Whether the intervention is delivered by a peer facilitator.
Period: Overall Study
Arm/Group | CD-LC | CBP- LC | QLW- LC | CD & CBP- LC | CD & QLW- LC | QLW & Capacity Building ProjectCBP- LC | QLW & CD & CBP-LC | Core LC | CD- PF | CBP- PF | QLW-PF | CD & CBP- PF | CD & QLW- PF | QLW & CBP- PF | CD & QLW & CBP- PF | Core PF
Started | 37 | 37 | 39 | 39 | 36 | 37 | 39 | 37 | 39 | 37 | 37 | 39 | 37 | 37 | 39 | 36
Completed | 14 | 24 | 27 | 32 | 26 | 17 | 30 | 30 | 26 | 26 | 26 | 30 | 25 | 29 | 35 | 28
Not Completed | 23 | 13 | 12 | 7 | 10 | 20 | 9 | 7 | 13 | 11 | 11 | 9 | 12 | 8 | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD-LC | CBP- LC | QLW- LC | CD & CBP- LC | CD & QLW- LC | QLW & Capacity Building ProjectCBP- LC | QLW & CD & CBP-LC | Core LC | CD- PF | CBP- PF | QLW-PF | CD & CBP- PF | CD & QLW- PF | QLW & CBP- PF | CD & QLW & CBP- PF | Core PF | Total
Number analyzed (Participants) | 37 | 37 | 39 | 39 | 36 | 37 | 39 | 37 | 39 | 37 | 37 | 39 | 37 | 37 | 39 | 36 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 37 | 39 | 37 | 35 | 37 | 37 | 37 | 39 | 36 | 37 | 38 | 37 | 37 | 38 | 36 | 594
  >=65 years | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 37 | 37 | 39 | 39 | 36 | 37 | 39 | 37 | 39 | 37 | 37 | 39 | 37 | 37 | 39 | 36 | 602
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 4 | 4 | 3 | 4 | 5 | 3 | 4 | 6 | 4 | 4 | 6 | 2 | 4 | 2 | 66
  Not Hispanic or Latino | 33 | 30 | 34 | 35 | 32 | 32 | 34 | 34 | 35 | 31 | 33 | 35 | 31 | 35 | 35 | 34 | 533
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 15
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 32 | 28 | 31 | 34 | 27 | 30 | 34 | 32 | 33 | 30 | 29 | 36 | 33 | 31 | 32 | 27 | 499
  White | 2 | 2 | 6 | 1 | 4 | 2 | 2 | 3 | 6 | 3 | 3 | 0 | 2 | 2 | 1 | 8 | 47
  More than one race | 2 | 5 | 0 | 1 | 2 | 3 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 3 | 3 | 0 | 27
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 8
Religion [Count of Participants; unit: Participants]
  Christian | 13 | 20 | 21 | 16 | 14 | 23 | 19 | 16 | 20 | 15 | 22 | 19 | 22 | 19 | 18 | 22 | 299
  Muslim | 14 | 9 | 4 | 11 | 11 | 5 | 14 | 14 | 7 | 7 | 9 | 8 | 7 | 11 | 12 | 7 | 150
  Other | 10 | 8 | 14 | 12 | 11 | 9 | 7 | 7 | 12 | 15 | 6 | 12 | 8 | 7 | 9 | 7 | 154
Sexual Preference/Orientation [Count of Participants; unit: Participants]
  Heterosexual | 34 | 36 | 37 | 33 | 33 | 30 | 34 | 33 | 32 | 36 | 31 | 34 | 35 | 35 | 36 | 33 | 542
  LGBTQ+ | 3 | 1 | 2 | 7 | 3 | 0 | 5 | 4 | 7 | 1 | 6 | 5 | 2 | 2 | 3 | 3 | 54
Marital Status [Count of Participants; unit: Participants]
  Married | 2 | 5 | 1 | 1 | 3 | 5 | 9 | 2 | 3 | 6 | 5 | 4 | 2 | 3 | 5 | 2 | 58
  Not married | 35 | 32 | 38 | 38 | 33 | 32 | 30 | 35 | 36 | 31 | 32 | 35 | 35 | 34 | 34 | 34 | 544
Employment status [Count of Participants; unit: Participants]
  Employed | 7 | 6 | 8 | 5 | 6 | 6 | 13 | 4 | 7 | 4 | 9 | 9 | 6 | 5 | 1 | 6 | 102
  Unemployed | 30 | 31 | 31 | 34 | 30 | 31 | 26 | 33 | 32 | 33 | 28 | 30 | 31 | 32 | 38 | 30 | 500
Substance Use [Mean (Standard Deviation); unit: %days past 30 days used substances] | 0.18 (0.12) | 0.24 (0.21) | 0.21 (0.16) | 0.18 (0.15) | 0.17 (0.15) | 0.23 (0.18) | 0.19 (0.19) | 0.19 (0.18) | 0.17 (0.13) | 0.24 (0.21) | 0.16 (0.16) | 0.20 (0.15) | 0.25 (0.16) | 0.21 (0.16) | 0.20 (0.13) | 0.17 (0.15) | 0.20 (0.16)
Time since release from Incarceration [Mean (Standard Deviation); unit: Years] | 5.36 (1.34) | 5.20 (1.26) | 4.95 (.83) | 5.75 (1.45) | 5.62 (1.74) | 5.08 (1.13) | 5.51 (1.44) | 5.85 (1.92) | 5.29 (1.50) | 5.65 (1.32) | 5.82 (2.70) | 5.00 (1.21) | 5.56 (1.31) | 5.53 (1.19) | 5.14 (1.18) | 5.61 (1.86) | 5.43 (1.52)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days of Alcohol or Substance Misuse in the Past 30 Days
Description: The primary outcome was the percentage of ASM (i.e., the percentage of days each substance was used in the past month) as operationalized by the Global Assessment of Individual needs. At each time point (baseline, five follow-ups), percentage ASM was calculated by dividing the reported number of days in the past month that participants used cannabis, heroin, alcohol, opioids, or cocaine by the number of days in the month (data were collected with the Timeline Follow-Back measure), multiplied by 100. Next, mean ASM frequency per month during 5 months of follow-up was calculated by adding the percentages for each substance and dividing by 5.31 We conducted correlations for self-reported ASM in the past 30 days with toxicology urine screens to assess validity of self-reported data.
Time Frame: 5 months
Population: Participants who completed 5 months post baseline follow-up
Measure: Mean (Standard Deviation); unit: % days misusing substances past 30 days
Arm/Group | CD-LC | CBP- LC | QLW- LC | CD & CBP- LC | CD & QLW- LC | QLW & Capacity Building ProjectCBP- LC | QLW & CD & CBP-LC | Core LC | CD- PF | CBP- PF | QLW-PF | CD & CBP- PF | CD & QLW- PF | QLW & CBP- PF | CD & QLW & CBP- PF | Core PF
Number analyzed (Participants) | 9 | 22 | 25 | 31 | 23 | 14 | 27 | 24 | 21 | 24 | 25 | 26 | 23 | 27 | 31 | 27
% days misusing substances past 30 days | 0.15 (0.12) | 0.16 (0.10) | 0.21 (0.12) | 0.16 (0.12) | 0.14 (0.11) | 0.22 (0.25) | 0.18 (0.13) | 0.17 (0.13) | 0.14 (0.15) | 0.21 (0.11) | 0.16 (0.12) | 0.15 (0.13) | 0.19 (0.12) | 0.14 (0.11) | 0.19 (0.16) | 0.14 (0.10)

2. Secondary Outcome: Number of People Abstinent From Alcohol and Drug Use
Description: Number of people abstinent from alcohol and drug use, which is assessed via the timeline follow back scale
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | CD-LC | CBP- LC | QLW- LC | CD & CBP- LC | CD & QLW- LC | QLW & Capacity Building ProjectCBP- LC | QLW & CD & CBP-LC | Core LC | CD- PF | CBP- PF | QLW-PF | CD & CBP- PF | CD & QLW- PF | QLW & CBP- PF | CD & QLW & CBP- PF | Core PF
Number analyzed (Participants) | 37 | 37 | 39 | 39 | 36 | 37 | 39 | 37 | 39 | 37 | 37 | 39 | 37 | 37 | 39 | 36
Participants | 1 | 1 | 0 | 2 | 3 | 0 | 1 | 3 | 4 | 2 | 3 | 4 | 0 | 7 | 3 | 5

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | CD-LC | CBP- LC | QLW- LC | CD & CBP- LC | CD & QLW- LC | QLW & Capacity Building ProjectCBP- LC | QLW & CD & CBP-LC | Core LC | CD- PF | CBP- PF | QLW-PF | CD & CBP- PF | CD & QLW- PF | QLW & CBP- PF | CD & QLW & CBP- PF | Core PF
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/39 | 0/39 | 0/36 | 0/37 | 0/39 | 0/37 | 0/39 | 0/37 | 0/37 | 0/39 | 0/37 | 0/37 | 0/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/39 | 0/39 | 0/36 | 0/37 | 0/39 | 0/37 | 0/39 | 0/37 | 0/37 | 0/39 | 0/37 | 0/37 | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/39 | 0/39 | 0/36 | 0/37 | 0/39 | 0/37 | 0/39 | 0/37 | 0/37 | 0/39 | 0/37 | 0/37 | 0/39 | 0/36

LIMITATIONS AND CAVEATS:
Only self-identified men were included in the study and it is critical to conduct comparable studies with people who identify with all genders. Further, future research is needed to replicate these findings and expand their generalizability to other regions, marginalised communities, and outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02951455/Prot_SAP_ICF_000.pdf